CLINICAL TRIAL: NCT05330039
Title: Enterobacteria Strain-level Characterization in Children With Inborn Errors of Metabolism (IEM)
Brief Title: Characterization of Intestinal Microbiota in Children With Inborn Errors of Metabolism (IEM)
Acronym: IEM
Status: Completed | Type: Observational
Sponsor: Emma Marie Caroline Slack (Other)
Collaborators: University Children's Hospital (Other)
Responsible Party: Sponsor-Investigator, Emma Marie Caroline Slack, Prof. Dr., ETH Zurich
Organization: ETH Zurich (Other)
Other Study IDs: IEM
Record Dates: First submitted 2022-03-31; First posted 2022-04-15 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Inborn Errors of Metabolism; Propionic Aciduria; Methylmalonic Aciduria; Urea Cycle Disorder
MeSH Terms: conditions — Metabolism, Inborn Errors; Propionic Acidemia; Methylmalonic acidemia; Urea Cycle Disorders, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with IEM: Collection of biological samples (stool and urine) and health-related data at two timepoints, three to six months apart.
- Healthy Siblings: Collection of biological samples (stool) and health-related data at two timepoints, three to six months apart.

SUMMARY:
Study around children with inborn errors of metabolism (IEM) and their healthy siblings. Collection of stool and urine to assess contribution of microbiota to disease severity.

DETAILED DESCRIPTION:
This study aims to collect biological samples (stool and urine) from children with inborn errors of metabolism, IEM (like UCD (urea cycle disorder), PA (propionic aciduria) and MMA (methylmalonic aciduria) and their healthy siblings.

The main focus of the study is to assess the contribution of the intestinal microbiota to disease severity in children that suffer from different forms of IEM and potentially find microbiota targets that could be used in the design of therapeutic/prophylactic agents.

ELIGIBILITY:
Inclusion Criteria:

* Children or siblings of children that have been diagnosed with one of the following diseases: any type of UCD, PA or MMA

Exclusion Criteria:

* Children or siblings of children that have not been diagnosed with one of the following diseases: any type of UCD, PA or MMA
* use of an investigational drug or device less than 30 days prior to the study, or current enrollment in another investigational drug or device study less than 30 days prior to the study
* considered to be poor attendees or unlikely for any reason to be able to comply with the study procedures, in the opinion of the investigator

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study aims to enroll 40 children that suffer from IEM (UCD, PA, MMA) and their siblings over the course of approximately two years.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-02-27 (Actual)

PRIMARY OUTCOMES:
Contribution of micriobiota to disease severity | 6 months
  Assess contribution of intestinal microbiota to disease severity in children that suffer from different forms of IEM via changes in frequencies, absolute colonization levels or strain identity of microbiota species

SECONDARY OUTCOMES:
Disease aggravating microbiota (microbiota target) | 6 months
  Identify members of the intestinal microbiota (species/strains) that are associated with IEM via differential abundance testing (microbiota target)

CONTACTS AND LOCATIONS:
Locations (1):
- University Children's Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No